CLINICAL TRIAL: NCT02206061
Title: School-based Asthma Care for Teens (SB-ACT)
Acronym: SB-ACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jill Halterman, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 51912; R18HL116244-01A1 (NIH)
Record Dates: First submitted 2014-07-25; First posted 2014-08-01 (Estimated); Results first posted 2021-02-21 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- School-Based Asthma Care for Teens (SB-ACT) (Experimental): SB-ACT consists of 2 components: Motivational Interviewing (MI) and Directly Observed Therapy (DOT) For the first 6-8 weeks, the teen will visit the school nurse to receive a daily dose of preventive asthma medication as directly observed therapy (DOT). The purpose of DOT is to establish a relationship with the nurse, learn proper medication technique, and experience potential benefits of consistent preventive therapy.
  The second component, Motivational Interviewing (MI) counseling , will start 4-6 weeks after the start of DOT. A counselor will conduct 3 in-person MI sessions with the teen at school to enhance the teen's motivation to adhere to their asthma treatment plan. The 3 sessions consist of an initial 40 minute counseling session (4-6 weeks after start of DOT), and two 30 minute follow-up sessions 2 and 6 weeks later. This component consists of an evidence-based self-management program to help the teen begin to transition to independence with preventive medication use.
  Interventions: Behavioral: School-Based Asthma Care for Teens (SB-ACT)
- Directly Observed Therapy (Active Comparator): For the first 6-8 weeks after enrollment, the teen will visit the school nurse once a day to receive a daily dose of preventive asthma medication as directly observed therapy (DOT).
  Interventions: Behavioral: Directly Observed Therapy
- Asthma Education (Active Comparator): Asthma educators will provide an in-school asthma education program that will match the time and attention of the MI counseling portion of the primary intervention. Each teen will receive three 1-on-1 educational sessions at school, and sessions will cover 3 main topics: 1) lung physiology and asthma basics, 2) triggers, symptoms, and warning signs, and 3) medications and self-advocacy.
  Interventions: Behavioral: Asthma Education

INTERVENTIONS:
Behavioral: School-Based Asthma Care for Teens (SB-ACT)
  Arms: School-Based Asthma Care for Teens (SB-ACT)
Behavioral: Directly Observed Therapy
  Arms: Directly Observed Therapy
Behavioral: Asthma Education
  Arms: Asthma Education

SUMMARY:
The goal of this study is to evaluate the widespread implementation of a developmentally appropriate preventive asthma care intervention for urban teens. The School Based Asthma Care for Teens (SB-ACT) program includes two core components: 1) a trial of directly observed therapy (DOT) to allow the teen to experience the potential benefits from adhering to guideline-based asthma treatment, and 2) a developmentally appropriate Motivational Interviewing (MI) Counseling Intervention to help the teen transition to independent long-term medication adherence. The investigators hypothesize that teens receiving the SB-ACT program will 1) experience less asthma-related morbidity than an asthma education (AE) attention-control comparison group, and 2) have improved adherence, less urgent healthcare use, less absenteeism, improved quality of life, and reduced FeNO compared to AE. The investigators also hypothesize that participants receiving DOT-only will have improved asthma-related outcomes immediately following their DOT trial vs. teens receiving AE, but will not have sustained, clinically significant improvement in outcomes once the DOT phase is complete. This represents a unique opportunity to build upon existing community relationships with an innovative and developmentally focused program to improve asthma outcomes for urban teens.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed asthma
* Persistent asthma or poor asthma control (based on NHLBI guidelines).
* Attending secondary school in Rochester City School District

Exclusion Criteria:

* Inability to speak and understand English
* No access to a phone for follow-up surveys
* Diagnosed developmental or intellectual disability
* Other significant medical conditions, including congenital heart disease, cystic fibrosis, or other chronic lung disease, that could interfere with the assessment of asthma-related measures.
* Teens in foster care or other situations in which consent cannot be obtained from a guardian.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 430 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2021-02-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Background] Frey SM, Fagnano M, Mammen JR, Halterman JS. Health-related internet use among adolescents with uncontrolled persistent asthma. J Asthma. 2021 Dec;58(12):1610-1615. doi: 10.1080/02770903.2020.1827420. Epub 2020 Oct 7. PMID 32969289
- [Background] Stern J, Chen M, Jusko TA, Fagnano M, Jarvinen KM, Halterman JS. Food allergy in at-risk adolescents with asthma: A key area for focus. Ann Allergy Asthma Immunol. 2020 Oct;125(4):405-409.e1. doi: 10.1016/j.anai.2020.06.004. Epub 2020 Jun 10. PMID 32534023
- [Background] Okelo SO, Bilderback AL, Fagnano M, Halterman JS. Validity of asthma disease direction, bother, and risk as self-reported asthma morbidity measures in urban teens. J Allergy Clin Immunol Pract. 2020 Mar;8(3):1129-1131.e2. doi: 10.1016/j.jaip.2019.09.026. Epub 2019 Oct 9. No abstract available. PMID 31605762
- [Background] Frey SM, Jones MR, Goldstein NPN, Fagnano M, Halterman JS. Comparing inhaled medications reported by adolescents with persistent asthma and their caregivers. J Asthma. 2020 Sep;57(9):999-1005. doi: 10.1080/02770903.2019.1631342. Epub 2019 Jul 2. PMID 31264485
- [Background] Shankar M, Fagnano M, Blaakman SW, Rhee H, Halterman JS. Depressive Symptoms Among Urban Adolescents with Asthma: A Focus for Providers. Acad Pediatr. 2019 Aug;19(6):608-614. doi: 10.1016/j.acap.2018.12.004. Epub 2018 Dec 20. PMID 30578922
- [Background] Jones MR, Frey SM, Riekert K, Fagnano M, Halterman JS. Transition Readiness for Talking With Providers in Urban Youth With Asthma: Associations With Medication Management. J Adolesc Health. 2019 Feb;64(2):265-271. doi: 10.1016/j.jadohealth.2018.08.026. Epub 2018 Oct 30. PMID 30389202
- [Background] Okelo SO, Bilderback AL, Fagnano M, Halterman JS. Validation of Asthma Control Assessment Among Urban Adolescents Using the Asthma Control and Communication Instrument. J Allergy Clin Immunol Pract. 2019 Mar;7(3):962-968.e1. doi: 10.1016/j.jaip.2018.10.001. Epub 2018 Oct 11. PMID 30317005
- [Background] Frey SM, Jones MR, Goldstein N, Riekert K, Fagnano M, Halterman JS. Knowledge of Inhaled Therapy and Responsibility for Asthma Management Among Young Teens With Uncontrolled Persistent Asthma. Acad Pediatr. 2018 Apr;18(3):317-323. doi: 10.1016/j.acap.2018.01.006. Epub 2018 Jan 31. PMID 29369804
- [Result] Halterman JS, Riekert KA, Fagnano M, Tremblay PJ, Blaakman SW, Tajon R, Wang H, Borrelli B. Effect of the School-Based Asthma Care for Teens (SB-ACT) program on asthma morbidity: a 3-arm randomized controlled trial. J Asthma. 2022 Mar;59(3):494-506. doi: 10.1080/02770903.2020.1856869. Epub 2021 Jan 8. PMID 33307900

RESULTS

PARTICIPANT FLOW:
Groups:
- School-Based Asthma Care for Teens (SB-ACT): SB-ACT consists of 2 components: Motivational Interviewing (MI) and Directly Observed Therapy (DOT) For the first 6-8 weeks, the teen will visit the school nurse to receive a daily dose of preventive asthma medication as directly observed therapy (DOT). The purpose of DOT is to establish a relationship with the nurse, learn proper medication technique, and experience potential benefits of consistent preventive therapy.
  The second component, Motivational Interviewing (MI) counseling , will start 4-6 weeks after the start of DOT. A counselor will conduct 3 in-person MI sessions with the teen at school to enhance the teen's motivation to adhere to their asthma treatment plan. The 3 sessions consist of an initial 40 minute counseling session (4-6 weeks after start of DOT), and two 30 minute follow-up sessions 2 and 6 weeks later. This component consists of an evidence-based self-management program to help the teen begin to transition to independence with preventive medication use.
  School-Based Asthma Care for Teens (SB-ACT)
- Directly Observed Therapy: For the first 6-8 weeks after enrollment, the teen will visit the school nurse once a day to receive a daily dose of preventive asthma medication as directly observed therapy (DOT).
  Directly Observed Therapy
- Asthma Education: Asthma educators will provide an in-school asthma education program that will match the time and attention of the MI counseling portion of the primary intervention. Each teen will receive three 1-on-1 educational sessions at school, and sessions will cover 3 main topics: 1) lung physiology and asthma basics, 2) triggers, symptoms, and warning signs, and 3) medications and self-advocacy.
  Asthma Education
Period: Overall Study
Arm/Group | School-Based Asthma Care for Teens (SB-ACT) | Directly Observed Therapy | Asthma Education
Started | 149 | 142 | 139
Completed | 131 | 128 | 118
Not Completed | 18 | 14 | 21
Not completed — Withdrawal by Subject | 4 | 7 | 1
Not completed — Lost to Follow-up | 14 | 7 | 20

BASELINE CHARACTERISTICS:
Population: Baseline data was collected for all enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | School-Based Asthma Care for Teens (SB-ACT) | Directly Observed Therapy | Asthma Education | Total
Number analyzed (Participants) | 149 | 142 | 139 | 430
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.4 (1.2) | 13.4 (1.2) | 13.5 (1.2) | 13.4 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 55 | 65 | 190
  Male | 79 | 87 | 74 | 240
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 102 | 92 | 97 | 291
  Not Hispanic or Latino | 47 | 50 | 42 | 139
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 1 | 3
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 82 | 78 | 79 | 239
  White | 5 | 7 | 10 | 22
  More than one race | 61 | 55 | 48 | 164
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 149 | 142 | 139 | 430

OUTCOME MEASURES:

1. Primary Outcome: Average Number of Days Without Asthma Symptoms (Symptom Free Days) During Post-intervention Follow-up Interviews (3, 5 and 7 Months)
Description: The primary outcome measure is asthma morbidity between groups. The investigators will measure asthma morbidity by looking at the average number of days without asthma symptoms (symptom free days) over 2 weeks, during the post-intervention follow-up assessments (3, 5 and 7 months post baseline).
  Symptom free days are defined as 24 hour periods of no asthma symptoms including, coughing, wheezing, tightness in the chest or shortness of breath.
  Reported data reflects the number of symptom free days over 2 weeks averaged across 3, 5, and 7 month post-intervention follow-up assessments.
Time Frame: Average number of symptom free days, over 2 weeks, averaged across 3, 5, and 7 month post-intervention follow-up assessments.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | School-Based Asthma Care for Teens (SB-ACT) | Directly Observed Therapy | Asthma Education
Number analyzed (Participants) | 131 | 128 | 118
Days | 11.5 (2.9) | 11.4 (2.9) | 11.6 (2.8)
Statistical Analysis 1: Comparison: School-Based Asthma Care for Teens (SB-ACT) vs Directly Observed Therapy vs Asthma Education; Test type: Other — Repeated measure analyses testing the overall treatment effect were performed by fitting the Generalized Estimating Equation (GEE) with SFD at the three follow-up time points (3, 5, 7 months) as the dependent variable and treatment as independent variable. Normal error and identity link was specified and standard error was calculated using Sandwich estimator. Baseline SFDs, poverty level, and the presence of smokers in the home were controlled in the regression model; p < .05, Regression, Linear; Mean Difference (Net) = .9, Standard Deviation 2.6

ADVERSE EVENTS:
Time Frame: 1 year
Description: n/a - definition does not differ
Arm/Group | School-Based Asthma Care for Teens (SB-ACT) | Directly Observed Therapy | Asthma Education
All-Cause Mortality (participants affected / at risk) | 0/149 | 0/142 | 0/139
Serious Adverse Events (participants affected / at risk) | 0/149 | 0/142 | 0/139
Other Adverse Events (participants affected / at risk) | 0/140 | 0/142 | 0/139

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT02206061/Prot_SAP_000.pdf